CLINICAL TRIAL: NCT04096131
Title: Influence of Cataract Surgery on Early DME: the DICAT-II Study
Brief Title: Influence of Cataract Surgery on Early DME The DICAT-II Study
Acronym: DICAT-II
Status: Completed | Type: Observational
Sponsor: European School of Advanced Studies in Ophthalmology (Other)
Responsible Party: Principal Investigator, Giacomo Panozzo, Scientific Studies Coordinator, European School of Advanced Studies in Ophthalmology
Other Study IDs: DICAT-II
Record Dates: First submitted 2019-09-09; First posted 2019-09-19 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Macular Edema; Cataract Senile; Surgery--Complications
Keywords: diabetic macular edema; cataract; surgery
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SURGERY: subjects with early DME undergoing cataract surgery
  Interventions: Procedure: cataract surgery
- OBSERVATION: subjects with early DME

INTERVENTIONS:
Procedure: cataract surgery — phacoemulsification
  Groups: SURGERY

SUMMARY:
To determine if cataract surgery may have an impact on the natural history of early DME (E-DME)

DETAILED DESCRIPTION:
Cataract surgery worsens preoperative DME, deserving an adequate pre and postoperative treatment. A large British study demonstrated that even eyes without preexisting edema are at risk of DME development after surgery according to the gravity of retinopathy. A new DME classification (the ESASO Classification of DME) defines a new category of DME, named early DME (E-DME) as follow: presence of small intraretinal cysts associated with well-recognizable and detectable inner retinal layers, ellipsoid zone (EZ) and external limiting membrane (ELM), with increase in central subfield thickness (CST) and/or macular volume (MV) less than 30% of maximum normal values.

Due to its undetectable or minimal impact on visual function, E-DME has not yet been studied, and retinologists usually restrict treatment to more advanced cases.

E-DME is the most frequent type of DME among the population undergoing cataract surgery, estimated by DICAT-I Study in 20.7% of the diabetic subjects, corresponding to 5.4% of the general population.

It has been demonstrated that cataract surgery has a negative impact both on diabetic eyes with no DME and in eyes with advanced DME. Even E-DME therefore probably worsens after surgery but there are no data on this matter.

Study Objective: to determine if cataract surgery may have an impact on the natural history of early DME (E-DME) Study Design: prospective multi-center observational case-control study

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be identified during the regular preoperative cataract examination. In the presence of a diabetic patient, an OCT scan will be performed (according to the protocol, see below).

Only eyes with E-DME will be eligible for the study.

Inclusion criteria may be one of the following:

1. Diabetic patients with bilateral E-DME and bilateral cataract. Both eyes will be enrolled: one eye will receive surgery at M4, the other at the end of follow up (M8) or later (gold candidate).
2. Diabetic patients with bilateral E-DME and cataract in just one eye (gold candidate). The eye with E-DME and no cataract may be already pseudophakic (surgery performed at least 18 months before) or with clear media.
3. Diabetic patients with E-DME and cataract in just one eye
4. Diabetic patients with cataract and no E-DME in the eye scheduled for surgery but E-DME in the other eye. Only the eye with E-DME will be enrolled.

Exclusion Criteria:

1. Past ocular surgery of any kind (except for cataract surgery) or ocular pathologies other than diabetic retinopathy.
2. Macular edema considered to be due to a cause other than diabetic macular edema.
3. OCT examination suggesting that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema. In the case of ERM, an OCT scan must be sent to the Coordinating Center for approval.
4. Any ocular pathology or ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema
5. History of any therapy (anti-VEGF treatment, focal/grid macular photocoagulation, intravitreous or peribulbar corticosteroids) for DME or diabetic retinopathy in the past 12 months.
6. History of YAG capsulotomy performed within two months before enrollment.
7. Aphakia.
8. Evidence of uncontrolled glaucoma.
9. Intraocular pressure must be <25 mmHg, with no more than one topical glaucoma medication.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Groups GROUP 1: Eyes with E-DME scheduled for cataract surgery GROUP 2: Control Group. Eyes with E-DME and clear media, non-significant cataract, pseudophakic (Group 2a: phakic; Group 2b: pseudophakic) or eyes with cataract scheduled for surgery after the end of follow up.
  Gold candidate: patient with bilateral E-DME and cataract in at least one eye.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Influence of cataract surgery on E-DME | 4 months
  Changes in central subfield thickness (CST) and/or macular volume (MV) measured by SD-OCT in eyes with E-DME during the first 4 months after cataract surgery (Group 1) compared to eyes with the same condition but without any surgical intervention (Group 2).
  Eyes in both groups developing a "significant worsening" of E-DME, defined as an increase of at least 50 microns in central subfield thickness (CST) or 0.5 mm3 in macular volume (MV) measured by SD-OCT will be withdrawn from the study to receive adequate therapeutic intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- ESASO Scientific Projects, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No